CLINICAL TRIAL: NCT00003782
Title: A Three-Arm Randomized Trial to Compare Adjuvant Adriamycin and Cyclophosphamide Followed by Taxotere (AC-T); Adriamycin and Taxotere (AT); and Adriamycin, Taxotere, and Cyclophosphamide (ATC) in Breast Cancer Patients With Positive Axillary Lymph Nodes
Brief Title: Combination Chemotherapy in Treating Women With Stage I, Stage II, or Stage IIIA (cT1-3, N0-1, M0) Breast Cancer and Positive Axillary Lymph Nodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-30; CDR0000066914
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Doxorubicin + Cyclophosphamide, then Docetaxel (Experimental): Doxorubicin + Cyclophosphamide, then Docetaxel
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin
- Arm 2: Doxorubicin + Docetaxel (Experimental): Doxorubicin + Docetaxel
  Interventions: Drug: docetaxel; Drug: doxorubicin
- Arm 3: Doxorubicin + Docetaxel + Cyclophosphamide (Experimental): Doxorubicin + Docetaxel + Cyclophosphamide
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin

INTERVENTIONS:
Drug: cyclophosphamide — Arm 1: 600 mg/m2 IV every 21 days for 4 cycles; Arm 3: 500 mg/m2 IV every 21 days for 4 cycles
  Arms: Arm 1: Doxorubicin + Cyclophosphamide, then Docetaxel; Arm 3: Doxorubicin + Docetaxel + Cyclophosphamide
Drug: docetaxel — Arm 1: 100 mg/m2 IV every 21 days for 4 cycles; Arms 2 and 3: 75 mg/m2 IV every 21 days for 4 cycles
  Other Names: Taxotere
Drug: doxorubicin — Arm 1: 60 mg/m2 IV every 21 days for 4 cycles; Arms 2 and 3: 50 mg/m2 IV every 21 days for 4 cycles
  Other Names: Adriamycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving combination chemotherapy after surgery may kill any tumor cells remaining following surgery. It is not yet known which regimen of combination chemotherapy is more effective in treating breast cancer with positive axillary lymph nodes.

PURPOSE: Randomized phase III trial to compare the effectiveness of different regimens of combination chemotherapy in treating women who have undergone surgery for stage I, stage II, or stage IIIA breast cancer with positive axillary lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of adjuvant doxorubicin, cyclophosphamide, and docetaxel given concurrently vs adjuvant doxorubicin and cyclophosphamide followed by docetaxel, in terms of overall survival and disease-free survival, of women with breast cancer and positive axillary lymph nodes.
* Compare the efficacy of adjuvant doxorubicin and docetaxel vs regimens containing cyclophosphamide in these patients.
* Compare the toxic effects of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens. (Quality of life substudy closed to accrual as of 7/20/01.)
* Compare the differences in amenorrhea in premenopausal women in each treatment arm and its relationship to symptoms, quality of life (quality of life substudy closed to accrual as of 7/20/01), disease-free survival, and overall survival.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, number of positive nodes (1-3 vs 4-9 vs at least 10), sequential tamoxifen or anastrozole administration (yes vs no), and type of prior surgery and radiotherapy plan (mastectomy with no local or regional radiotherapy vs mastectomy with local and/or regional radiotherapy vs lumpectomy with local radiotherapy vs lumpectomy with local and regional radiotherapy). Patients are randomized to one of three treatment arms.

* Arm 1: Patients receive doxorubicin IV over 15 minutes and cyclophosphamide IV over 30 minutes every 21 days for 4 courses. Three weeks after the last dose of this combination, patients receive docetaxel IV over 1 hour every 21 days for 4 courses.
* Arm 2: Patients receive doxorubicin IV over 15 minutes and docetaxel IV over 1 hour every 21 days for 4 courses.
* Arm 3: Patients receive doxorubicin IV over 15 minutes, cyclophosphamide IV over 30 minutes, and docetaxel IV over 1 hour every 21 days for 4 courses.

Patients in all arms who are estrogen receptor-positive and/or progesterone receptor-positive receive oral tamoxifen daily for 5 years beginning within 3-12 weeks of completion of chemotherapy. Patients who are postmenopausal may receive alternative hormonal therapy at the discretion of the treating physician.

Some patients may receive postmastectomy radiotherapy on SWOG-S9927 or NCIC-MA.20 after recovery from chemotherapy.

Quality of life and menstrual history are assessed before randomization, on day 1 of course 4, and at 6, 12, 18, and 24 months. (Quality of life substudy closed to accrual as of 7/20/01.)

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 5,300 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive adenocarcinoma of the breast

  * Confined to the breast and ipsilateral axilla on clinical exam

    * Stage I, II, or IIIA (cT1-3, N0-1, M0)
* At least one axillary lymph node with evidence of tumor on histologic exam

  * Sentinel node biopsy allowed if followed by axillary dissection
  * No suspicious palpable nodes in the contralateral axilla or palpable supraclavicular or infraclavicular nodes, unless proven on biopsy to not be involved with tumor
* No bilateral malignancy or mass in the opposite breast, unless mass is histologically proven to be benign
* Must have undergone either a prior total mastectomy and axillary dissection (modified radical mastectomy) OR
* Prior lumpectomy and axillary dissection

  * Patients must receive radiotherapy after randomization (not before) AND after chemotherapy
  * Margins must be clear
  * No ipsilateral lymph nodes that are fixed to one another or to other structures (N2 disease) and/or any positive nonaxillary lymph nodes (intramammary nodes are considered axillary nodes)
  * No histologically evident invasive tumor or ductal carcinoma in situ
  * No diffuse tumors by mammography that would not be surgically amenable to lumpectomy
  * No other dominant mass in the ipsilateral breast remnant unless one of the following is true:

    * Histologically benign
    * Surgically removed with clear margins if malignant
* No ulceration, erythema, infiltration of the skin or underlying chest wall (complete fixation), peau d'orange, or skin edema of any magnitude

  * Tethering or dimpling of the skin or nipple inversion allowed
* No metastatic disease

  * Skeletal pain allowed if bone scan negative for metastases
* Hormone receptor status:

  * Estrogen and progesterone status determined

PATIENT CHARACTERISTICS:

Age:

* greater than or equal to 18 years

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* At least 10 years, excluding diagnosis of cancer

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3 (may be less, if in the opinion of the investigator, this represents an ethnic or racial variation)
* Platelet count at least 100,000/mm^3* NOTE: *If platelet count is above the upper limit of normal (ULN), significant underlying hematologic disorders must be excluded

Hepatic:

* Bilirubin no greater than ULN
* Alkaline phosphatase less than 2.5 times ULN*
* SGOT less than 1.5 times ULN*
* No nonmalignant systemic hepatic disease that would preclude study participation NOTE: *Alkaline phosphatase and SGOT cannot both be greater than ULN

Renal:

* Creatinine no greater than normal
* No nonmalignant systemic renal disease that would preclude study participation

Cardiovascular:

* No nonmalignant systemic cardiovascular disease that would preclude study participation
* LVEF at least lower limit of normal (LLN) by MUGA or echocardiogram
* No active cardiac disease that would preclude use of doxorubicin or docetaxel, including the following:

  * Any prior myocardial infarction
  * Angina pectoris requiring anti-anginal medication
  * History of congestive heart failure
  * Cardiac arrhythmia requiring medication
  * Severe conduction abnormality
  * Valvular disease with documented cardiac function compromise
  * Cardiomegaly on chest x-ray or ventricular hypertrophy on EKG, unless LVEF at least LLN
  * Poorly controlled hypertension (diastolic greater than 100 mm/Hg)
  * Hypertension well controlled by medication allowed

Other:

* No grade 2 or greater peripheral neuropathy
* No other prior malignancy within the past 5 years except:

  * Effectively treated squamous cell or basal cell skin cancer
  * Surgically treated carcinoma in situ of the cervix
  * Segmentally resected lobular carcinoma in situ of the ipsilateral or contralateral breast
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No nonmalignant systemic disease that would preclude study participation
* No diabetes with morning fasting blood glucose of 200 mg/dL or greater
* No psychiatric or addictive disorders that would preclude informed consent
* No contraindication to corticosteroids that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for breast cancer

Chemotherapy:

* No prior chemotherapy for breast cancer
* No prior anthracyclines or taxanes
* No other concurrent investigational chemotherapy

Endocrine therapy:

* No prior hormonal therapy for breast cancer
* No concurrent hormonal birth control methods or other hormonal therapy
* No concurrent raloxifene, including for osteoporosis
* Concurrent low-dose topical estrogen in the form of conjugated estrogen ring or conjugated estrogen vaginal cream (dose no more than 0.3 mg or 1/8 of an applicator applied vaginally 3 times a week) allowed

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy for this malignancy

Surgery:

* See Disease Characteristics
* No more than 84 days since prior surgery for breast cancer (e.g., lumpectomy, mastectomy, sentinel node biopsy, axillary dissection, or re-excision of lumpectomy margins)

Other:

* No prior systemic therapy for this malignancy
* No concurrent medications that alter cardiac conduction (e.g., digitalis, beta blockers, or calcium-channel blockers) for cardiac arrhythmia, angina, or congestive heart failure (allowed if administered for other reasons [e.g., hypertension])
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5351 (Actual)
Dates: Start 1999-03; Primary Completion 2008-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (157):
- United States (146):
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center, Fresno, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Scripps Cancer Center at Scripps Clinic, La Jolla, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Pacific Shores Medical Group, Long Beach, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Stanford Cancer Center at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Catholic Healthcare West - Westbay Region, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - University of Connecticut Cancer Center at University of Connecticut Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Norton Healthcare Cancer Center, Louisville, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Stanley S. Scott Cancer Center at Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C. - Albany Regional Cancer Center, Albany, New York
  - Charles R. Wood Foundation Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Staten Island University Hospital, Staten Island, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - Alamance Cancer Center, Burlington, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Jewish Hospital of Cincinnati, Incorporated, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - South Pointe Hospital - Cancer Care Center, Warrensville Heights, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baptist Cancer Institute - Memphis at Baptist Memorial Hospital - Memphis, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Virginia Oncology Associates - Newport News, Newport News, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (11):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec

REFERENCES:
- [Result] Swain SM, Land SR, Ritter MW, Costantino JP, Cecchini RS, Mamounas EP, Wolmark N, Ganz PA. Amenorrhea in premenopausal women on the doxorubicin-and-cyclophosphamide-followed-by-docetaxel arm of NSABP B-30 trial. Breast Cancer Res Treat. 2009 Jan;113(2):315-20. doi: 10.1007/s10549-008-9937-0. Epub 2008 Feb 27. PMID 18302020
- [Result] Ganz PA, Land SR, Geyer CE, et al.: NSABP B-30: definitive analysis of quality of life (QOL) and menstrual history (MH) outcomes from a randomized trial evaluating different schedules and combinations of adjuvant therapy containing doxorubicin, docetaxel and cyclophosphamide in women with operable, node-positive breast cancer. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-76, 2008.
- [Result] Swain SM, Jeong JH, Geyer CE, et al.: NSABP B-30: definitive analysis of patient outcome from a randomized trial evaluating different schedules and combinations of adjuvant therapy containing doxorubicin, docetaxel and cyclophosphamide in women with operable, node-positive breast cancer. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-75, 2008.
- [Result] Swain SM, Land SR, Sundry R, et al.: Amenorrhea in premenopausal women on the doxorubicin (A) and cyclophosphamide (C) followed-by docetaxel (T) arm of NSABP B-30: preliminary results. [Abstract] J Clin Oncol 23 (Suppl 16): A-537, 13s, 2005.
- [Derived] Bandos H, Melnikow J, Rivera DR, Swain SM, Sturtz K, Fehrenbacher L, Wade JL 3rd, Brufsky AM, Julian TB, Margolese RG, McCarron EC, Ganz PA. Long-term Peripheral Neuropathy in Breast Cancer Patients Treated With Adjuvant Chemotherapy: NRG Oncology/NSABP B-30. J Natl Cancer Inst. 2018 Feb 1;110(2):djx162. doi: 10.1093/jnci/djx162. PMID 28954297
- [Derived] Swain SM, Jeong JH, Geyer CE Jr, Costantino JP, Pajon ER, Fehrenbacher L, Atkins JN, Polikoff J, Vogel VG, Erban JK, Rastogi P, Livingston RB, Perez EA, Mamounas EP, Land SR, Ganz PA, Wolmark N. Longer therapy, iatrogenic amenorrhea, and survival in early breast cancer. N Engl J Med. 2010 Jun 3;362(22):2053-65. doi: 10.1056/NEJMoa0909638. PMID 20519679

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Doxorubicin + Cyclophosphamide, Then Docetaxel | Arm 2: Doxorubicin + Docetaxel | Arm 3: Doxorubicin + Docetaxel + Cyclophosphamide
Started | 1783 | 1784 | 1784
Completed | 1753 | 1753 | 1758
Not Completed | 30 | 31 | 26
Not completed — No follow up data | 30 | 31 | 26

BASELINE CHARACTERISTICS:
Groups:
- Doxorubicin + Cyclophosphamide, Then Docetaxel: Doxorubicin + Cyclophosphamide, then Docetaxel
- Doxorubicin + Docetaxel: Doxorubicin + Docetaxel
- Doxorubicin + Docetaxel + Cyclophosphamide: Doxorubicin + Docetaxel + Cyclophosphamide
- Total: Total of all reporting groups
Arm/Group | Doxorubicin + Cyclophosphamide, Then Docetaxel | Doxorubicin + Docetaxel | Doxorubicin + Docetaxel + Cyclophosphamide | Total
Number analyzed (Participants) | 1783 | 1784 | 1784 | 5351
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (9.8) | 50 (9.5) | 51 (9.9) | 51 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1783 | 1784 | 1784 | 5351
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: 8 years
Measure: Number; unit: percentage of patients alive
Arm/Group | Arm 1: Doxorubicin + Cyclophosphamide, Then Docetaxel | Arm 2: Doxorubicin + Docetaxel | Arm 3: Doxorubicin + Docetaxel + Cyclophosphamide
Number analyzed (Participants) | 1753 | 1753 | 1758
percentage of patients alive | 83 | 79 | 79

2. Primary Outcome: Disease Free Survival
Time Frame: time to event: breast cancer recurrence; second primary cancer; death from any cause as a first event
Reporting Status: Not Posted

3. Secondary Outcome: Toxicities Among the 3 Regimens
Time Frame: 9 years
Reporting Status: Not Posted

4. Secondary Outcome: Quality of Life Among Breast Cancer Patients
Time Frame: baseline, 9 weeks, and 6, 12, 18, and 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Amenorrhea in Premenopausal Women
Time Frame: baseline, 9 weeks, and 6, 12, 18, and 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Arm/Group | Doxorubicin + Cyclophosphamide, Then Docetaxel | Doxorubicin + Docetaxel | Doxorubicin + Docetaxel + Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 66/1748 | 43/1748 | 46/1745
Other Adverse Events (participants affected / at risk) | 845/1748 | 561/1748 | 641/1745
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin + Cyclophosphamide, Then Docetaxel (N=1748) | Doxorubicin + Docetaxel (N=1748) | Doxorubicin + Docetaxel + Cyclophosphamide (N=1745)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alanine aminotransferase increased (ALT/SGPT) (Investigations) | 1 | 0 | 1
Anaphylaxis (Immune system disorders) | 1 | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Aspartate aminotransferase increased (AST/SGOT) (Investigations) | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 3 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1 | 2
Conduction disorder (Cardiac disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 2 | 0 | 0
Creatinine increased (Investigations) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2
Depression (Psychiatric disorders) | 5 | 6 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 3
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 7
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 5 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 9 | 7 | 10
Intracranial hemorrhage (Nervous system disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 4 | 2
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Psychosis (Psychiatric disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 12 | 4 | 8
Typhlitis (Gastrointestinal disorders) | 1 | 3 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Wound infection (Infections and infestations) | 1 | 1 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0
Visceral arterial ischemia (Vascular disorders) | 0 | 0 | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin + Cyclophosphamide, Then Docetaxel (N=1748) | Doxorubicin + Docetaxel (N=1748) | Doxorubicin + Docetaxel + Cyclophosphamide (N=1745)
Arthralgia (Musculoskeletal and connective tissue disorders) | 126 | 22 | 33
Diarrhea (Gastrointestinal disorders) | 78 | 66 | 111
Fatigue (General disorders) | 212 | 135 | 167
Febrile neutropenia (Blood and lymphatic system disorders) | 383 | 223 | 275
Infections and infestations - Other, specify (Infections and infestations) | 200 | 144 | 137
Myalgia (Musculoskeletal and connective tissue disorders) | 148 | 29 | 35
Nausea (Gastrointestinal disorders) | 162 | 127 | 155
Vomiting (Gastrointestinal disorders) | 140 | 90 | 119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days